CLINICAL TRIAL: NCT05613595
Title: Effectiveness of Positive Psychotherapy on Mental Wellbeing, Sense of Coherence, Social Support and Difficulties Among Caregivers of Cerebral Palsy Children
Brief Title: Effectiveness of Positive Psychotherapy on Mental Wellbeing Among Caregivers of Cerebral Palsy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Islamic University, Islamabad (Other)
Responsible Party: Principal Investigator, Saima Waqar, Principal Investigator, International Islamic University, Islamabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60-FSS/PHDPSY/F18
Record Dates: First submitted 2022-10-28; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Caregiver Burden; Mental Health Issue; Cerebral Palsy
Keywords: Positive psychotherapy; Sense of Coherence; Social support
MeSH Terms: conditions — Caregiver Burden; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Present study will be conducted on caregivers of Cerebral palsy children. It will be conducted in four phases. In phase I, Urdu translation & adaptation of Caregiver Difficulties Scale (CDS) and Positive Psychotherapy (PPT) manual will be done. .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychotherapy Group (Active Comparator): In this phase of the study, the caregivers of CP having moderate to high scores on mental health issues on three scales (Depression, Burnout & Caregiver burden) will receive positive Psychotherapy sessions for a period of four months, divided over different weekly sessions. For Psychotherapy treatment group participants will be given both counseling as well as Positive psychotherapy based interventions. . Each session will be based upon individual session and duration of the session will be 40 minutes. Before starting every session feedback will be taken about the previous session and home based assignments will also be discussed
  Interventions: Behavioral: Positive Psychotherapy
- Counseling Group (Active Comparator): 10 participants will be included in in control group (N=10), for control group caregivers will be given regular counseling as a part of treatment of their child (psychoeducation). Each session will be based upon individual session and duration of the session will be 40 minutes.
  Interventions: Behavioral: Counseling Group

INTERVENTIONS:
Behavioral: Positive Psychotherapy — Positive Psychotherapy is an effective treatment for many mental disorders and depression is primary empirical target. Its primary goal is to build positive emotion, engagement, and meaning in life that will alleviate depression and other mental health disorders. Thus PPT may offer a new way to treat and prevent mental health issues.
  Interventions sessions included, Session Records Session One: Positive Introduction and Gratitude Journal Session Two: Character Strengths and Signature Strengths Session Three: Practical Wisdom , Session Four: A Better Version of Me , Session Five: Open and Closed Memories, Session Six: Forgiveness Session Seven: Maximizing versus Satisficing, Session Eight: Gratitude ,Session Nine: Hope and Optimism, Session Ten: Posttraumatic Growth, Session Eleven: Slowness and Savoring, Session Twelve: Positive Relationships, Session Thirteen: Positive Communication, Session Fourteen: Altruism , Session Fifteen: Meaning and Purpose
  Arms: Positive Psychotherapy Group
Behavioral: Counseling Group — Caregivers in control group only regular counseling will be provided (psychoeducation). it will be based upon the insight of cerebral palsy and training based on Adaptive skill functioning of the CP child of the caregivers
  Arms: Counseling Group

SUMMARY:
The Central idea of the proposed research proposal is first to translate adapt and validate the Caregiver Difficulties Scale & Positive Psychotherapy sessions based manual into Urdu language then secondly, assessment of burnout, burden, depression, mental wellbeing, sense of coherence and social support among caregivers of Cerebral palsy children and finally measuring the effectiveness of Positive Psychotherapy for treating mental health issues of caregivers of Cerebral Palsy children. This research proposal will provide an Urdu language based standardized positive psycho therapeutic based intervention to mental health practitioners for treating mental health issues of caregivers of cerebral palsy children in sociocultural context of Pakistan. In Pakistan earlier conducted researches mainly focused on assessment of mental health issues of caregivers of cerebral palsy children, however present research will not only assess the sample regarding their mental health issues, but in addition it will also contribute in provision of psychometrically sound Urdu language based positive Psychotherapy. Positive Psychotherapy focuses on positive emotions and personal strengths instead of ruminating over weaknesses.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a congenital neurodevelopmental disorder, due to non-progressive disability it prolongs throughout ages. Mental health of the caregivers of CP children is affected due to prolong treatment of the child. Keeping in mind the long term multiple disability in cerebral palsy much focus in earlier researches were given to the rehabilitation of the child and less attention is given to address the mental health issues of caregivers of cerebral palsy children. The current study is based on identifying the mental health issues like depression, caregiver burden and burnout among caregivers of CP children and how sense of coherence and social support have impact on the mental wellbeing of caregivers of CP children. After measuring the level of mental health issues of care givers of cerebral palsy children, the present study also aimed at rehabilitation of the caregivers of cerebral palsy children with the help of positive psychotherapy in rehabilitation unit. The positive psychotherapy based interventions will be translated and adapted in Urdu language for the present study. According to the literature review no such positive psychotherapy based techniques used on caregivers of CP Children in Pakistan. Positive Psychotherapy is selected as an interventional therapy in the present study and for the first time it has been planned for this sample in Pakistan. Core focus of positive psychotherapy is to move away the client from negative aspect of life and focus them towards the positive aspects of life. If positive psychotherapy treatment is effective as compared to traditional treatment approach it will be cost effective and will reduce caregiver burden, depression and burnout.

ELIGIBILITY:
Inclusion Criteria:

* Only those participants will be included who would have moderate to high score on caregiver burden, depression & burnout and lower score in wellbeing, social support & sense of coherence.

Interventions will be given to the caregivers having moderate level of burnout & depression.

Inclusion Criteria

* Caregiver will be someone who takes the primary responsibility for caregiving a child with CP.
* Only caregivers of Diagnosed CP child
* Caregivers having only 1 CP child in the family
* Educational status of the care giver will be matric and above.
* Age of CP child under 10 years Exclusion Criteria:• Caregivers with any severe diagnosed Psychiatric illness (psychosis & depressive Illness) will not be added in the present study.
* More than 1 CP child in the family
* Caregivers who are Uneducated will not be added in the present study.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-01-12 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Parental Burnout Assessment | baseline and 8th week
  a 23- item self-report questionnaire for assessment of Burn Out
Change in Depression Anxiety Stress Scale | baseline and 8th week
  DASS is a self-report 21 items based questionnaire designed to measure depression, anxiety and stress
Change in Caregiver Difficulties Scale | baseline and 8th week
  a self-administered questionnaire measure the caregiver burden
Change in Sense of Coherence | baseline and 8th week
  Measured by the orientation of life scale, It contains 13 items
Change in wellbeing Positive Psychotherapy Inventory | baseline and 8th week
  self-report inventory having 25 items.it assess level of mental wellbeing,
Change Multidimensional Scale of Perceived Social Support | baseline and 8th week
  Social support is measured across three domains; friends, family and significant others. The responses reflect participant's perception of support from each of these three sources

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Mushtaq, PhD, Study Director — International Islamic University, Islamabad
Locations (1):
- National Institute of Rehabilitation Medicine, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No